CLINICAL TRIAL: NCT06353841
Title: The Effect of Therapeutic Touch on Functional Constipation in Infants and Young Children: A Randomized Controlled Study
Brief Title: Effect of Therapeutic Touch on Functional Constipation in Infants and Young Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Burdur Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Selda Ateş Beşirik, Principal Investigator, Burdur Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/435
Record Dates: First submitted 2024-03-31; First posted 2024-04-09 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Functional Constipation; Therapeutic Touch; Infants; Children; Constipation
Keywords: Therapeutic Touch; Functional Constipation; Infants; Children
MeSH Terms: conditions — Constipation | interventions — Therapeutic Touch

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The data analyst will be blinded to the procedure and results of randomization, group allocation, and intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Therapeutic Touch will be applied to infants for three consecutive days, once a day, ten minutes at any time during the day. There will be a four-day break. The Therapeutic Touch will be done a total of three times in one week.
  Interventions: Behavioral: Therapeutic Touch
- Control group (No Intervention): The therapeutic touch will not be applied to the control group infants.

INTERVENTIONS:
Behavioral: Therapeutic Touch — Therapeutic Touch will be applied to infants for 3 consecutive days, once a day, 10 minutes at any time during the day. There will be a four-day break. The Therapeutic Touch will be done a total of 3 times a week in four weeks.
  Arms: Intervention Group

SUMMARY:
The aim of the study is to determine the effect of therapeutic touch on functional constipation in infants and young children.

DETAILED DESCRIPTION:
Functional constipation (FK) is a common functional gastrointestinal disorder that affects children's quality of life. The reported prevalence of functional constipation in infants and young children varies according to diagnostic criteria between studies. Laxatives and probiotics are commonly used to treat functional constipation. Therefore, treating constipation is very costly and there is not enough reliable data on this subject. When the literature is examined, the use of non-pharmacological methods to reduce, prevent and eliminate constipation has been increasing recently. When the studies were examined, studies using different methods were found. The main methods used in the care of children with constipation are; massage, aromatherapy, probiotics, laxatives, reflexology and acupuncture. The effect of therapeutic touch is thought to have positive results, especially in newborns, infants and children.Based on the studies conducted in line with the literature, this research has a randomized controlled experimental design to determine the effect of therapeutic touch applied to infants and children diagnosed with functional constipation according to Rome IV criteria on constipation.

This study is a prospective, randomized and controlled trial. The study population consisted of infants and children aged 6 to 24 months. Sample of the study consisted of a total of 60 children who met the sample selection criteria and were selected via randomization method. Children were randomized into two groups: intervention gorup (n=30) and control group (n=30). Data were collected using the Interview and Observation Form, Primary Results Follow-up Form, and Bristol stool form scale.

ELIGIBILITY:
Inclusion Criteria:

* The infant is between 6-24 months,
* The infant was born at term,
* Birth weight between 2500-4500 g,
* Must have been diagnosed with functional constipation by the physician according to ROMA IV criteria,
* Mothers' ability to read, write and speak Turkish,
* Parent's willingness to participate in the research.

Exclusion Criteria:

* The infant has a congenital anomaly,
* The infant has any chronic disease,
* Having a secondary disease that causes constipation such as cow's milk allergy, celiac disease, hypercalcemia and hypothyroidism, neurological diseases,Children with any organic or metabolic diseases
* The parent has a verbal and written communication barrier.

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2024-12-26 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Primary Results Follow-up Form | In four weeks
  Weekly Bowel sounds (movements) (min)
Primary Results Follow-up Form | In four weeks
  Number of stools
Primary Results Follow-up Form | In four weeks
  Stool density
Primary Results Follow-up Form | In four weeks
  Weight (g)
Primary Results Follow-up Form | In four weeks
  Abdominal circumference (cm)

SECONDARY OUTCOMES:
Bristol Stool Scale | In four weeks
  In this scoring system, stool hardness is evaluated from the hardest to the softest, according to the adhesion and cracking characteristics of the stool.
  In this scoring system, stool hardness is from the hardest to the softest, according to the adhesion and cracking characteristics of the stool; is divided into seven classes: hard scattered tubers like hazelnuts:Type 1, sausage-shaped but lumpy:Type 2, like a sausage but with cracks on the surface:Type 3, smooth and soft like a sausage or snake:Type 4, soft grains with obvious cuts on the edges:Type 5, mushy stool with irregular edges and fluid pieces:Type 6, watery, with no solid pieces, and completely liquid:Type 7. Type 1 and Type 2 are difficult defecation patterns and suggest the presence of constipation, Type 3, Type 4 and Type 5 indicate normal defecation, and Type 6 and Type 7 suggest diarrhea.
Constipation discomfort | In four weeks
  Child's Distress Intensity: The child's discomfiture intensity during defecation will be defined. (0-3 points: "0" no crying or grimace, "1" mild crying and grimace, "2" moderate crying and grimace, "3" hysterical intense crying and grimace.) (Zhang et al., 2022).

CONTACTS AND LOCATIONS:
Overall Officials: Selda Ateş Beşirik, PhD., Principal Investigator — Burdur Mehmet Akif Ersoy University; Emine Geçkil, Professor, Study Director — Necmettin Erbakan University
Locations (1):
- Burdur Bucak State Hospital, Burdur, Bucak, Turkey (Türkiye)